CLINICAL TRIAL: NCT06840301
Title: The Effect of Mindfulness Compassionate Living Training on Ruminative Thinking and Sleep Quality in Informal Caregivers of Inpatients in Palliative Clinic: a Randomized Controlled Trial
Brief Title: The Effect of Mindfulness Compassionate Living Training on Ruminative Thinking and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mine CENGİZ, Lecturer Physician, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCENGİZ4
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Mindfulness Compassionate Living Training
Keywords: Mindfulness; Sleep Quality; Ruminative Thinking
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Session 1: How We Evolved - Threat, Impulse, and Soothing Systems (Experimental): * A "breath break with kindness" is practiced.
  * Encourage them to think about how threat, impulse and sedative systems have developed in their own lives.
  * A "safe place" application is made.
  * "Courtesy meditation" is done.
  Interventions: Behavioral: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems
- Session 2: Threat and Self-Compassion (Experimental): * A "breath break with kindness" is practiced.
  * "Building a compassionate relationship with resilience" and "kindness meditation: a benevolent" practices are made.
  * "A hand on your heart" and "a compassionate comrade" practices are made.
  Interventions: Behavioral: Session 2: Threat and Self-Compassion
- Session 3: Unraveling the Knots of Desire and Patterns Agenda (Experimental): * Talk about homework.
  * A "breath break with kindness" is practiced.
  * "Establishing a compassionate relationship with desire", "guided meditation to discover the inner pattern", "courtesy meditation: a good friend" practices are made.
  Interventions: Behavioral: Session 3: Unraveling the Knots of Desire and Patterns
- Session 4: Internalizing compassion (Experimental): * "Pretend-to-pretend" practice is made for participants to observe themselves.
  * In addition to the previous practices, the practice of "internalizing compassion" is made in order to increase their expanded mindfulness.
  * Courtesy meditation: a neutral person", "kindness towards your body", which is based on mindfulness practices and increases body awareness and mindful movement, is carried out.
  During the day, they will be informed that they should do the "walking with kindness" practice on their own.
  Interventions: Behavioral: Session 4: Internalizing compassion
- Session 5: Me and others - Expanding the circle (Experimental): * A "compassionate letter" application is made by asking participants to think about a situation they encountered recently or some time ago and is still causing distress. It is explained that they can gain insight with this application.
  * "Courtesy meditation: the 'difficult' person", "compassion and breathing: yourself" and "compassionate breathing: others" practices are made
  Interventions: Behavioral: Session 5: Me and others - Expanding the circle
- Session 6: Growing happiness (Experimental): * "Revisiting the good" practice is carried out to define the five sense organs for the participants.
  * "Forgiveness", "Asking for forgiveness", "forgiving others", "gratitude" practices are carried out.
  * The practice is expanded as "kindness meditation: groups and all beings".
  Interventions: Behavioral: Session 6: Growing happiness
- Session 7: Weaving Wisdom and Compassion into Daily Life (Experimental): * Participants are made to choose a day in their life and allow a few minutes to pause in a mindful way.
  * "A breather for wise and compassionate action", "calmness meditation" and "joy sharing meditation" practices are carried out.
  Interventions: Behavioral: Session 7: Weaving Wisdom and Compassion into Daily Life
- Session 8: Living with the Heart (Experimental): * The participants are told about the applications that they can apply for, where they need help to develop compassion towards self-healing skills, and the whole training is evaluated.
  * The "river of life" application, which evaluates mindfulness in depth, is carried out.
  * An overall summary of the 8-session study is made and feedback is received.
  Interventions: Behavioral: Session 8: Living with the Heart

INTERVENTIONS:
Behavioral: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems — The practice of "Breath break with kindness" will be applied for 5 minutes. Afterwards, 15 minutes of information on threats, impulses and soothing systems, "A safe place" application for 11 minutes, "Courtesy meditation" for 10 minutes. After each application, 10 minutes of feedback will be received from the participants.
  Arms: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems
Behavioral: Session 2: Threat and Self-Compassion — The practice of "breathing with kindness" will be done for 7 minutes. The practice of "Building a compassionate relationship with resilience" will be held for 12 minutes, and the practice of "Kindness meditation: a benevolent" will take place for 11 minutes. "A hand over your heart" application will be made for 3 minutes and "A compassionate comrade" application will be done for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 2: Threat and Self-Compassion
Behavioral: Session 3: Unraveling the Knots of Desire and Patterns — The practice of "breathing with kindness" will be done for 7 minutes. "Building a compassionate relationship with desire" 12 minutes, "Guided meditation to discover the inner pattern" 10 minutes and "Courtesy meditation: a good friend" 11 minutes. Except for the "breath break with kindness" application, 3 minutes of feedback will be received from the participants after each application
  Arms: Session 3: Unraveling the Knots of Desire and Patterns Agenda
Behavioral: Session 4: Internalizing compassion — The "pretend-to-be" practice for the participants to observe themselves will be made for 10 minutes. The practice of "internalizing compassion" will be done for 7 minutes, "kindness meditation: a neutral person" practice for 10 minutes, and "kindness towards your body" for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 4: Internalizing compassion
Behavioral: Session 5: Me and others - Expanding the circle — The "a compassionate letter" practice with the participants will continue for 15 minutes. "meditation: the 'difficult' person" 8 minutes, "compassion and breathing: yourself" 10 minutes and "compassionate breathing: others" 7 minutes. A "compassionate break" application is performed for 7 minutes.
  Arms: Session 5: Me and others - Expanding the circle
Behavioral: Session 6: Growing happiness — The practice of "Revisiting the good" is carried out for 10 minutes with the participants. "Forgive yourself", "wish for forgiveness", "forgive others", "gratitude" practices will be held for 5 minutes each and will take 20 minutes in total. "Courtesy meditation: groups and all beings" will be practiced for 10 minutes. After each application, 3 minutes of feedback will be received from the participants
  Arms: Session 6: Growing happiness
Behavioral: Session 7: Weaving Wisdom and Compassion into Daily Life — Participants will be given 10 minutes to choose a day in their life and allow a few minutes to pause mindfully. The practice of "a breather for wise and compassionate action" is 10 minutes, the practice of "calmness meditation" is 8 minutes, and the practice of "sharing the joy meditation" is 8 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 7: Weaving Wisdom and Compassion into Daily Life
Behavioral: Session 8: Living with the Heart — The participants are told about the applications they can apply for, where they need help to develop compassion towards self-healing skills, and the entire training will be evaluated for 20 minutes. The "river of life" application is carried out for 20 minutes. 10 minutes of feedback will be received after the application.
  Arms: Session 8: Living with the Heart

SUMMARY:
This study was planned to evaluate the effects of Mindfulness Compassionate Living training on ruminative thinking and sleep quality in informal caregivers of patients in a palliative clinic in Turkey. The data of the study will be conducted between November 2024 and April 2025 in the Palliative Clinic of Atatürk University Health Research and Application Center located in the city center of Erzurum. The universe of the study will consist of individuals between the ages of 18 and 45 who are caregivers of patients in the palliative clinic during the specified date range. The sample size of the study was calculated using the GPower computer program. In the calculation made with the power analysis at α=0.05 level, the effect size was 150, 153 (d=0.8) and the power of the study was 90%, it was calculated that at least 68 patients should be included in the sample. Patients who meet the research criteria and agree to participate in the study will be randomly assigned to one experimental and one control group.An introductory information form prepared by the researcher in line with the literature, containing the socio-demographic data of patients and their caregivers in the palliative clinic, the Ruminative Thinking Style Scale to assess the general thought tendency of individuals, the Level 2 Sleep Disorder Adult Short Form (PROMIS) to assess sleep quality, the Self-Compassion Scale Short Form (SCI-S) to assess self-compassion, and the Mindful Awareness Scale (MMIS) to assess conscious awareness will be used.

DETAILED DESCRIPTION:
Research data will be collected face to face by the researcher. The study will be conducted with informal caregivers who meet the inclusion criteria (being a caregiver of the patient in a palliative clinic, being willing to participate in the research, being open to communication and cooperation). Pre-test measurement tools will be applied to the informal caregivers participating in the study. Then, Mindfulness Compassionate Living Training will be applied. Eight After the session application process, the final test data will be applied.

ELIGIBILITY:
Inclusion Criteria:

1. Being a caregiver of a patient in a palliative clinic,
2. Being between the ages of 18 and 45,
3. Being willing to participate in the study
4. Being open to communication and cooperation

Exclusion Criteria:

1. Having a psychiatric problem in the caregiver of a patient in a palliative clinic.
2. Not being open to communication and cooperation,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | up to 1 day
  The form consists of 16 questions prepared by the researcher within the scope of the literature, including information about the patient and caregiver in the palliative clinic. The created form includes questions covering the caregiver's age, gender, place of residence, education status, social security, marital status, profession and the process in which he/she provided care to the patient.

SECONDARY OUTCOMES:
Ruminative Thinking Style Scale | up to 1 day
  The scale developed by Brinker and Dozois ignores the individual's current feelings and moods and tries to understand the general tendency of thought. This scale can also be used in other pathological conditions. The Ruminative Thinking Style Scale has a 7-point Likert-type scoring system ranging from 1 to 7, with 1 being "not descriptive at all" and 7 being "describes me very well". In this scale, participants indicate to what extent the statements in the scale reflect themselves by scoring options from 1 to 7. The Turkish version of this scale was carried out in our country by Karatepe, Yavuz and Türkcan; the Cronbach Alpha coefficient of the scale was found to be 0.90.

OTHER OUTCOMES:
Level 2 Adult Sleep Disorder Short Form (PROMIS) | up to 1 day
  Sleep disturbance will be assessed using the Patient Reported Outcome Measurement Information System (PROMIS®) Short Form - Sleep Disorder. All seven items will be rated on a 5-point scale ranging from "Very poor" to "Very good" for the first item and from "Not at all" to "Very much" for all other items. Item 2 of the scale is reverse coded.
Self-Compassion Scale Short Form (SCI-K) | up to 1 day
  The scale developed by Neff (2003) was validated and reliable in Turkish by Yıldırım and Sarı in 2018. The scale was confirmed to have a structure consisting of 11 items, a single dimension, and two complementary components (positive component and negative component). The internal consistency coefficient of the scale was calculated as .75. It is recommended that it be used in studies where the total score will be used to measure self-compassion.
Conscious Awareness Scale (CAS) | up to 1 day
  It was developed by Brown and Ryan27 for the purpose of evaluating the BF level of individuals. In the validity and reliability study of the scale conducted in a university sample in Turkey, the Cronbach alpha coefficient was determined as 0.80.28 The scale is a one-dimensional, six-point Likert-type scale consisting of 15 questions. The minimum and maximum scores that individuals can get from the scale are between 15 and 90. High scores indicate a high BF level.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Tosun Taşar (Associate Professor), Study Chair — Ataturk University Faculty of Medicine
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided